CLINICAL TRIAL: NCT04256330
Title: Cardiometabolic Health and Inflammatory Resolution (Kardiometabol hälsa Och Inflammatorisk Resolution)
Brief Title: Cardiometabolic Health and Inflammatory Resolution
Acronym: REX
Status: Recruiting | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-04179
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Lean and metabolically healthy
- Lean and metabolically unhealthy
- Overweight and metabolically healthy
- Overweight and metabolically unhealthy
- Obese and metabolically healthy
- Obese and metabolically unhealthy

SUMMARY:
The aim of this study is to determine how inflammatory resolution impacts cardiometabolic health and disease in subjects that are either lean (18.5-24.9 kg/m2), overweight (25.0-29.9 kg/m2) or obese (>30.0 kg/m2).

ELIGIBILITY:
Inclusion Criteria:

* Informed signed consent has been obtained from the volunteer.
* The volunteer has a BMI greater than 18.5 kg/m2

Exclusion Criteria:

* The study staff contacting a potential participant perceives that the individual has difficulty understanding the information.
* An MD determines that the individual is on too many medications to participate
* The individual takes a medication that is approved by the MD, but he/she is not willing or not able to wait with any potential morning medication until after their fasted blood-draw.
* The individual is younger than 18 years (relevant for the FAINT-1 and FAINT-2 cohorts)
* The individual states that they have increased bleeding tendency or are using anti-coagulant (blood thinning) medication.
* The individual has some form of chronic inflammation.
* The individual regularly uses medication that affects inflammatory resolution (e.g., low-dose aspirin).
* The individual uses immunosuppressive drugs (eg, methotrexate).
* The individual regularly consumes fish oils (omega 3).
* The individual has significant gastrointestinal problems.
* The individual smokes or uses chewing tobacco.
* The individual has been drinking alcohol two days before the study visit.
* The individual has tattoos or body piercings on the forearms and / or the stomach that can affect the examination.
* The individual does not follow instructions given in the research study.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects are recruited either via open adds of after having indicated in previous study registers that they are interested in participating as volunteers in future studies.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Inflammatory status | 2027
  The inflammatory status, defined as CRP levels and ability to respond to pro-resolving therapeutics, will be studied in all 6 groups

CONTACTS AND LOCATIONS:
Locations (1):
- Gothenburg university, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No